CLINICAL TRIAL: NCT05916976
Title: MRI in Repaired Tetralogy of Fallot: Risc Score Derived From Multiparametric Magnetic Resonance-Imaging and Clinical Data to Sharpen the Indication for Change of Individualized Treatment
Brief Title: Repaired Tetralogy of Fallot: Risc Score From MRI & Clinical Data to Predict the Need for Change of Treatment
Acronym: rTOF-MR-SHARP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Joachim Lotz, Professor of Radiology; Director Institute of Diagnostic and Interventional Radiology, University Medical Center Goettingen
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-02659
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Tetralogy of Fallot; Congenital Heart Disease
Keywords: MRI; Tetralogy of Fallot; Multiparametric score; cardiac
MeSH Terms: conditions — Tetralogy of Fallot; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: all patients scheduled for MRI for follow-up of repaired Tetralogy of Fallot.
Masking Description: MRI data are made available for clinical decision. Score will not be made available to treatment decision team. Nor is the study team involved in the clinical decision process until completion of follow-up data acquisition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rTOF-patients (Other): rTOF-patients with age 16 and above enrolled in Adult Congenital Heart Disease (ACHD)-outpatient clinics program with regularly scheduled MRI-exam
  Interventions: Diagnostic Test: cardiac MRI

INTERVENTIONS:
Diagnostic Test: cardiac MRI — Multiparametric MRI of the heart

SUMMARY:
Patient with Tetralogy of Fallot need live-long surveillance after initial operative correction (rTOF). MRI is an established and important component of the standardized follow-up in this patient population. A new score will be used to summarize the multitude of MRI-based parameters into a single number. Individual modificators are assigned to the components of the score. The value of each modificatory will be determined as a result of this feasibility trial. This new compound score is designed to anticipate any deterioration of cardiac function, arrhythmias or sudden cardiac death. This feasibility study is the first step to establish this score and find initial values for the modifies that are assigned to the more than 40 biomarkers from MRI, clinical examinations and serum parameters that are included in this new score.

DETAILED DESCRIPTION:
Patient with Tetralogy of Fallot need live-long surveillance after initial operative correction (rTOF). MRI is an established and important component of the standardized follow-up in this patient population. Though a large number of diverse MRI-derived parameter have been shown to correlate with the incidence of major adverse cardiac events in patients with rTOF, there is not a single MRI-derived parameter that reliably predicts the incidence of heart failure, malignant arrhythmias or sudden cardiac death - the most common major adverse cardiac events in this group (rTOF-MACE). This feasibility trial is set to evaluate the feasibility of a weighted compound risk score based on about 40 parameters derived from MRI and augmented by clinical as well as serum-based biomarkers. This trial will recruit 70 consecutive patients with rTOF and correlate the new compound score with the clinical course over 2 years and the incidence of any change in therapy due to cardiac reasons. At the end of the trial each of the contributing parameters of the compound score will have been assigned a modifier based on its statistical relevance for the prediction of patient-specific rTOF-MACE or any change in cardiac related therapy. Based on this feasibility trial we aim to use the weighted compound score in a large multicenter trial to proof its applicability and relevance to short, medium and longterm prognosis of this special patient group.

ELIGIBILITY:
Inclusion Criteria:

* rTOF; age above 16; eligible for MRI-exam

Exclusion Criteria:

* any contraindications to MRI; unstable patient; unresponsive patient

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Modified therapy cardiovascular | 24 months
  Any change in therapy related to cardiovascular function

SECONDARY OUTCOMES:
hospitalization | 24 months
  Need of hospital admission due to any cardiovascular cause
cardiac intervention | 24 months
  Any cardiac invasive / minimal invasive intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Lotz, MD, Study Director — Institute of Diagnostic and Interventional Radiology, UMG Göttingen
Locations (1):
- University Medical Center Goettingen, Göttingen, Lower Saxxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
Results of all successfully included patients, anonymized.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After completion of study and publication of results. probably 2026
Access Criteria: Access granted upon qualified request. Data will be made available through the RACOON Network of the Network of University Medicine Germany (NUM-Project) as well as the German Center of Cardiovascular Research (DZHK)